CLINICAL TRIAL: NCT03848416
Title: Relative Bioavailability of 2 Ixekizumab Test Formulations Compared to the Commercial Formulation in Healthy Subjects
Brief Title: A Study of Ixekizumab in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 17140; I1F-MC-RHCT (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Results first posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-01

CONDITIONS: Healthy
MeSH Terms: interventions — ixekizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ixekizumab (Reference) (Experimental): Reference formulation ixekizumab 80 milligram (mg) administered as a subcutaneous (SC) injection in a prefilled syringe.
  Interventions: Biological: Ixekizumab
- Ixekizumab (Test 1) (Experimental): Test 1 formulation ixekizumab 80 mg administered as an SC injection in a prefilled syringe.
  Interventions: Biological: Ixekizumab
- Ixekizumab (Test 2) (Experimental): Test 2 formulation ixekizumab 80 mg administered as an SC injection in a prefilled syringe.
  Interventions: Biological: Ixekizumab

INTERVENTIONS:
Biological: Ixekizumab — Administered SC
  Other Names: LY2439821

SUMMARY:
The purpose of this study is to compare three different formulations of ixekizumab. One formulation (Reference) has been approved by the Food and Drug Administration (FDA) and two formulations (Test 1 and Test 2) have not been approved. This study will compare how much of each of the three formulations get into the blood stream. Information about any side effects that may occur will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participant or female participant who agree to not become pregnant
* Are male participant or female participants with chronic stable medical problems, that in the investigator's opinion will not place the subject at increased risk by participating in the study

Exclusion Criteria:

* Have a significant history of, or current, cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, or hematologic disorders that in the opinion of the investigator poses an unacceptable risk to the participant if participating in the study
* Are allergic or hypersensitive to the study medicine
* Had a vaccination with a live vaccine within 12 months prior to the first check-in or intend to get a vaccine for tuberculosis within 12 months of completing treatment on this study
* Have any type of hepatitis, human immunodeficiency virus (HIV) infection, or other serious infection
* Show evidence of active or latent tuberculosis (TB)
* Presence of significant neuropsychiatric disorder or a recent history of depression
* Have had any active or recent infection within 4 weeks of Day 1 that, in the opinion of the investigator would pose an unacceptable risk to the participant, if participating in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Inc, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to 1 of 3 treatments, Reference, Test Formulation 1 or Test Formulation 2.
Period: Overall Study
Arm/Group | Ixekizumab (Reference) | Ixekizumab (Test 1) | Ixekizumab (Test 2)
Started | 33 | 33 | 33
Received at Least One Dose of Study Drug | 33 | 33 | 33
Completed | 32 | 33 | 32
Not Completed | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Ixekizumab (Reference): Reference formulation ixekizumab 80 mg administered as a subcutaneous (SC) injection in a prefilled syringe.
- Total: Total of all reporting groups
Arm/Group | Ixekizumab (Reference) | Ixekizumab (Test 1) | Ixekizumab (Test 2) | Total
Number analyzed (Participants) | 33 | 33 | 33 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (13.5) | 41.9 (15.9) | 49.2 (15.2) | 44.5 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 24 | 69
  Male | 11 | 10 | 9 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 11 | 11 | 36
  Not Hispanic or Latino | 19 | 22 | 22 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 7 | 6 | 20
  White | 25 | 25 | 27 | 77
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 33 | 33 | 99

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Ixekizumab
Description: Pharmacokinetics (PK): Maximum Concentration (Cmax) of a single dose of Ixekizumab
Time Frame: Predose, Day 3, Day 5, Day 11, Day 15, Day 22, Day 29, Day 36, Day 43, Day 57, Day 71 and Day 85 Post Dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (ug/mL)
Arm/Group | Ixekizumab (Reference) | Ixekizumab (Test 1) | Ixekizumab (Test 2)
Number analyzed (Participants) | 33 | 33 | 33
microgram/milliliter (ug/mL) | 6.31 (48) | 6.29 (33) | 6.50 (33)

2. Primary Outcome: PK: Area Under the Plasma Concentration Versus Time Curve (AUC) From Time Zero to the Last Measured Concentration Value (AUC[0-tlast]) of Ixekizumab
Description: Area under the plasma concentration versus time curve from time zero to the last measured concentration value (AUC[0-tlast]). AUC 0-tlast is equal to AUC (0-85) days where the last time point was 85 Days ± 3 Days.
Time Frame: Predose, Day 3, Day 5, Day 11, Day 15, Day 22, Day 29, Day 36, Day 43, Day 57, Day 71 and Day 85 Post Dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day/milliliter (ug*day/mL)
Arm/Group | Ixekizumab (Reference) | Ixekizumab (Test 1) | Ixekizumab (Test 2)
Number analyzed (Participants) | 32 | 33 | 32
microgram*day/milliliter (ug*day/mL) | 146 (43) | 153 (37) | 163 (33)

3. Primary Outcome: PK: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Ixekizumab.
Description: Area under the plasma concentration versus time curve from zero to infinity (AUC[0-∞]) of a single dose of Ixekizumab.
Time Frame: Predose, Day 3, Day 5, Day 11, Day 15, Day 22, Day 29, Day 36, Day 43, Day 57, Day 71 and Day 85 Post Dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*day/mL
Arm/Group | Ixekizumab (Reference) | Ixekizumab (Test 1) | Ixekizumab (Test 2)
Number analyzed (Participants) | 32 | 33 | 32
ug*day/mL | 152 (45) | 159 (38) | 170 (34)

ADVERSE EVENTS:
Time Frame: Up to 12 Weeks
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Ixekizumab (Reference) | Ixekizumab (Test 1) | Ixekizumab (Test 2)
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33 | 1/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 1/33
Other Adverse Events (participants affected / at risk) | 4/33 | 2/33 | 5/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixekizumab (Reference) (N=33) | Ixekizumab (Test 1) (N=33) | Ixekizumab (Test 2) (N=33)
Periorbital abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Phaeohyphomycotic brain abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cerebral venous thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixekizumab (Reference) (N=33) | Ixekizumab (Test 1) (N=33) | Ixekizumab (Test 2) (N=33)
Injection site reaction (General disorders) | 1 (1) | 2 (2) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT03848416/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/16/NCT03848416/SAP_001.pdf